CLINICAL TRIAL: NCT07065201
Title: Effectiveness of a Digital prE-operative patieNt guIdance systeM (DENIM) in Enhancing Preparation of Elective Patients Undergoing Anesthesia: a Randomized Controlled Trial
Brief Title: DENIM-trial: Digital prE-operative patieNt guIdance systeM
Acronym: DENIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeroen Bosch Ziekenhuis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2022.04.04.02
Record Dates: First submitted 2025-06-24; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Rate of Late Cancellation; Patient Adherence to Preoperative Instructions; Patient Satisfaction; Care Givers Satisfaction
Keywords: patient guidance; mobile application; digital support; late cancellations; adherence; preoperative instructions; satisfaction
MeSH Terms: conditions — Patient Satisfaction; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: single center randomized trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in the intervention arm are individuals scheduled for elective surgery who will be asked to download a mobile application specifically designed for preoperative guidance. Through this app they will receive all relevant preoperative instructions via automated reminders and push notifications (e.g., fasting, medication adjustment). In addition, they will be asked to complete a short questionnaire via the app.
  Interventions: Device: Mobile application for preoperative patient guidance
- Control group (Placebo Comparator): Patients in the control group are individuals scheduled for elective surgery who will be asked to download the same mobile application as the intervention group. However, they will not receive any preoperative instructions through the app. They will be asked to fill out the same questionnaire as the control group.
  Interventions: Device: Mobile application and standard care

INTERVENTIONS:
Device: Mobile application for preoperative patient guidance — The mobile application provides patients with tailored information during the preoperative period until seven days after surgery. 1) Before the preoperative outpatient clinic visits, patient will receive information regarding the preoperative screening process and an overview of available anesthesia techniques through videos embedded in the app. 2) After approval for surgery and during the period leading up to the day of surgery, they will receive instructions concerning medication adjustment, lifestyle modifications, fasting rules, and hygiene measures.
  Arms: Intervention group
Device: Mobile application and standard care — Patients in the control group will be asked to download the same mobile app but they will not receive the same tailored information as those in the intervention group. Instead, they will be provided with standard preoperative information and instructions. In addition, they will be asked to fill out the same questionnaire as the intervention group.
  Arms: Control group

SUMMARY:
The goal of this RCT is to assess the effectiveness of a mobile application in enhancing the preoperative preparation of patients scheduled for elective surgery under anesthesia or procedural sedation. The main object is to evaluate the effect of preoperative instructions, delivered through reminders and push notifications, on the rate of late cancellations. Secondary outcomes are adherence to preoperative instructions, patient satisfaction, and care provider satisfaction.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of two groups: 1) Intervention group: patients will be asked to download a mobile application specifically designed for preoperative guidance. Through this app they will receive all relevant preoperative instructions via automated reminders and push notifications (e.g., fasting and medication adjustment). In addition, they will be asked to complete a short questionnaire via the app. 2) Control group: patients will download the same mobile application and will be asked to fill out the same questionnaire. However, they will not receive any preoperative instructions through the app. All patients in both groups will continue to receive the standard written instructions. App access will be maintained until five days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* patients scheduled for elective surgery under anesthesia or procedural sedation
* Possession of a mobile phone or tablet
* Access to a valid email address for study communication

Exclusion Criteria:

* age < 18 years
* emergency surgery
* language barrier
* no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Rate of late cancellations | Day of surgery
  Unexpected cancellation of a scheduled surgical case on the day of surgery, prior to the procedure taking place.

SECONDARY OUTCOMES:
Adherence to preoperative instructions | Day of surgery
  Adherence to instruction regarding anticoagulants, antihypertensive medication, hypoglicaemic medication, astma/COPD medication, fasting rules. This outcome will be assessed as a binary outcome (yes/no) based on wether the patients has followed all relevant preoperative instructions.
Patient satisfaction | 7 days after surgery
  Patient satisfaction will be assessed using the Usability: System Usability Scale (SUS)/ Mobile App Usability Questionnaire (MAUQ)1. Vaarious aspects of the app's use will be evaluated including quality, quantity and timing of information provided. Satisfaction will be measured on a numerical scale from 0 (not satisfied at all) to 10 (extremely satisfied).
Care provider satisfaction | At 6 and 12 months after implementation
  preoperative screening nurses and surgeons will be asked to complete a questionnaire at 6 and 12 months after implementation. Their experince with patient's use of the app will be assessed using a numerical rating scale ranging from 0 (not usefull at all) to 10 (extremely usefull)

CONTACTS AND LOCATIONS:
Locations (1):
- Jeroen Bosch Hospital, 's-Hertogenbosch, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
No plan made yet